CLINICAL TRIAL: NCT02281669
Title: Prospective Observational Study of Intralesional Treatment With Pentostam in Cutaneous Leishmaniasis Israeli Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Prof. Eli Schwartz MD, DTMH, Principal investigator of the geographic clinic, Sheba medical center, Sheba Medical Center
Other Study IDs: SHEBA-14-1571-ES-CTIL
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-10

CONDITIONS: Cutaneous Leishmaniasis
MeSH Terms: conditions — Leishmaniasis, Cutaneous | interventions — Antimony Sodium Gluconate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Research group: The study group includes all CL cases for whom the treating physician decides to treat by IL Pentostam. The patients will return to follow up and additional treatment every 3 weeks until full recovery [as our current policy].
  Interventions: Drug: Pentostam

INTERVENTIONS:
Drug: Pentostam — Intralesional injection of Pentostam
  Other Names: Pentavalent antimonials

SUMMARY:
Cutaneous leishmaniasis (CL) is endemic in Israel and is caused by Leishmania major or Leishmania tropica. CL is usually a benign disease and limited to the skin. One of the local treatment available is intralesional (IL) Pentostam injection. During the current study the investigators will monitor the adverse effects of this treatment and will follow up the recovery of the lesions after Pentostam injections.

DETAILED DESCRIPTION:
Cutaneous leishmaniasis is usually treated by topical intervention. In more severe cases intralesional Pentostam injection may be applied. This treatment is extremely efficient but painful, however without the known adverse effects of IV Pentostam treatment.

In this study the investigators will follow systematically all leishmania patients who are receiving the intralesional treatment. A structured questionnaire will be filled up in each doctor visit.

The current study goal is to examine the adverse effects and the patient reaction to this treatment, and to follow the recovery of lesion(s) after this treatment including the number of IL injections which was needed.

ELIGIBILITY:
Inclusion Criteria:

* Cutaneous leishmaniasis patients
* Treatment by IL Pentostam
* Age above 18 years

Exclusion Criteria:

* Children and pregnant women will not participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients arriving to the Geographic clinic or to the Skin clinic, diagnosed with Cutaneous leishmaniasis, and the treatment which is choosen by their physican is Pentostam injections.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2016-11 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Adverse effects | 1 year
  The adverse effects of IL Pentostam treatment will be monitored during the follow up period.

SECONDARY OUTCOMES:
Lesion healing | 1 year
  Lesions number and size will be recorded and response to treatment will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Schwartz, M.D, DTMH, Principal Investigator — Sheba Medical Center
Locations (1):
- Center of Geographic Medicine, Tel Litwinsky, Israel